CLINICAL TRIAL: NCT03740100
Title: Open-label, Single Arm, Two-stage Study, Evaluating the Efficacy and Safety of Bimiralisib in Patients With Recurrent or Metastatic Head and Neck Squamous Cell Carcinomas (HNSCC) Harboring NOTCH1 Loss of Function (LOF) Mutations
Brief Title: Single-arm Study With Bimiralisib in Patients With HNSCC Harboring NOTCH1 Loss of Function Mutations
Acronym: HNSCC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was closed because the sponsor became insolvent.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-1003 (PQR309-009); NCI-2019-02978 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2018-11-01; First posted 2018-11-14 (Actual); Results first posted 2022-01-20 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: HNSCC
Keywords: Head and Neck Squamous Cell Carcinoma; Notch 1 loss of function mutation; PI3K/mTOR Inhibitor; Refractory metastatic
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Oral administration
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open single arm (Other): Bimiralisib capsules orally
  Interventions: Drug: Bimiralisib

INTERVENTIONS:
Drug: Bimiralisib — Bimiralisib capsules
  Other Names: PQR309, PI3K/mTOR inhibitor

SUMMARY:
Preclinical data and limited clinical evidence suggest that Head and Neck Squameous Cell Carcinoma tumors harboring certain mutations may respond well to PI3K/mTOR inhibition (phosphatidylinositol-3-kinase/ mammalian target of rapamycin inhibition).

The current study enrolls patients with refractory and / or metastatic Head and Neck Squameous Cell Carcinoma based on the mutational status of their disease to assess the response to treatment with bimiralisib, an orally available pan-PI3K/mTOR inhibitor (phosphatidylinositol-3-kinase/ mammalian target of rapamycin inhibitor).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytological confirmed diagnosis of Head and Neck Squameous Cell Carcinoma, for which no standard curative or life prolonging therapy is available
2. Available CLIA-certified sequencing results of the NOTCH gene in Head and Neck Squameous Cell Carcinoma (HNSCC) tumor material. The tumor must harbor a NOTCH1 LOF mutation as confirmed by central review (MD Anderson Cancer Center, MDACC)
3. ECOG performance status of ≤ 2
4. Adequate bone marrow, liver, and renal functions
5. Measurable disease according to RECIST version 1.1
6. Patients of reproductive potential must agree to use effective contraception from screening until 90 days after discontinuing study treatment.

Exclusion Criteria:

1. Has received any anti-cancer treatment including hormonal and investigational agents within 21 days prior to first dose of bimiralisib.
2. Major surgery within 28 days prior to first dose of bimiralisib or persisting side effects that have not improved to NCI-CTCAE grade 1 or better.
3. Pregnant or nursing (lactating) women.
4. Poorly controlled diabetes mellitus, steroid-induced diabetes mellitus
5. Has other active malignancies that require systemic treatment.
6. Has a known history of HIV infection
7. Any of the following cardiac abnormalities:

   * History of, or current, documented congestive heart failure (New York heart association functional classification iii - iv), documented cardiomyopathy
   * Symptomatic (NYHA class II or higher) left ventricular ejection fraction (LVEF) < 40% as determined by multiple gated acquisition (MUGA) scan or echocardiogram (echo)
   * Myocardial infarction ≤ 6 months prior to enrolment
   * Unstable angina pectoris
   * Serious uncontrolled cardiac arrhythmia
   * Symptomatic pericarditis
8. Impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug.
9. Patient has a history of non-compliance to medical regimen or inability to grant consent.
10. Medically documented history of an active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others) or ≥ CTCAE grade 3 anxiety
11. History of interstitial pneumonitis or patients who require chronic oxygen supplementation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Faye M Johnson, MD,PhD, Principal Investigator — MD Anderson Cancer Center Recruiting, Houston, Texas, US 77030
Locations (1):
- M.D. Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Johnson FM, Janku F, Gouda MA, Tran HT, Kawedia JD, Schmitz D, Streefkerk H, Lee JJ, Andersen CR, Deng D, Rawal S, Shah PA, El-Naggar AK, Johnson JM, Frederick MJ. Inhibition of the Phosphatidylinositol-3 Kinase Pathway Using Bimiralisib in Loss-of-Function NOTCH1-Mutant Head and Neck Cancer. Oncologist. 2022 Dec 9;27(12):1004-e926. doi: 10.1093/oncolo/oyac185. PMID 36124629
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Bimilralisib: Bimiralisib capsules orally.
  All patients received 140 mg bimiralisib (PQR309) 140 mg orally once daily on two consecutive days followed by five days without treatment weekly until unacceptable toxicity, tumor progression, patient's request for withdrawal, investigator judgment, or death.
Period: Overall Study
Arm/Group | Bimilralisib
Started | 8 (Note: Ten patients were consented, but two died before starting therapy.)
Confirmed Partial Response | 1 (Using a Simon's optimal two-stage design, we planned to enroll up to 10 evaluable patients in the first stage. Two of eight treated patients were not evaluable for response based on toxicity. We did not reach this milestone.)
Completed | 6
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- Bimiralisib Treatment: Bimiralisib capsules (140 mg) orally once daily on 2 consecutive days followed by 5 days without treatment weekly.
Arm/Group | Bimiralisib Treatment
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 65.5 [50 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Radiological tumor assessments were performed by computed tomography (CT) or magnetic resonance imaging (MRI) according to a standard protocol.
  ORR: comprised of all patients who achieved a confirmed partial or a confirmed complete response per RECIST 1.1
Time Frame: At 6 and 12 weeks after the start of therapy (± 3 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Open Single Arm
Number analyzed (Participants) | 6
Participants | 1
Statistical Analysis 1: Comparison: Open Single Arm; The primary endpoint was to determine the objective response rate of patients with R/M HNSCC harboring NOTCH1 LOF mutations to oral bimiralisib using RECIST v1.1. We used a Simon's optimal two-stage design. In order to have 80% power to detect a response rate of 30%, (one-sided α=0.05 and β=0.20), we planned to enroll up to 10 patients in the first stage. If ≥ 2 patients had an objective response, then the study would enroll an additional 19 patients in the second stage; Test type: Other; Percent with objective response = 17, 95% CI 2-sided [1 to 58]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug (bimiralisib) until 30 days after the last dose of bimiralisib.
Arm/Group | Open Single Arm
All-Cause Mortality (participants affected / at risk) | 2/8
Serious Adverse Events (participants affected / at risk) | 5/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Single Arm (N=8)
Disease Progression (General disorders) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Hyperglycemia (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal Stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal Injury (Renal and urinary disorders) | 1 (1)
Hemorrhage (Vascular disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Single Arm (N=8)
Platelet count decreased (Blood and lymphatic system disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Blood creatinine increased (Renal and urinary disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
vomiting (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 2 (3)
Tinnitus (Ear and labyrinth disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial was closed early because the sponsor became insolvent.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT03740100/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT03740100/SAP_001.pdf
  • Informed Consent Form (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT03740100/ICF_002.pdf